CLINICAL TRIAL: NCT03165162
Title: Assessing Consumer's Characterization of the Term Natural in a Food Context
Acronym: NTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB2017-042
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: natural; Food Label Choices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Food Order: Randomly assigned orders of 7 bowls of granola, each with a different food label.
  Interventions: Behavioral: Food Order

INTERVENTIONS:
Behavioral: Food Order — randomly assigned orders of 7 bowls of granola, each with a different food label.

SUMMARY:
The purpose of this project is to gain a better understanding of the underlying consumer motivations associated with choosing foods labeled as "natural"; and further, how the use of this term impacts the amount of food consumed.

DETAILED DESCRIPTION:
This study is a randomized, 1-arm, parallel trial design focused on determining the types of food labels people associate with 'natural.' A planned sample size of 100 will be enrolled into the study. This study will require one initial screening visit and 1 Study Day. This study will take approximately 1 day to 1 week per subject to complete.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, and exercise habits.

If willing and eligible to participate, subjects will be invited to participate in the study for 1 Study Day that participants can choose to continue on to after the Screening visit.

Subject will arrive at the center in a fasted. During the Study Day, each participant will be asked to complete a health and mindfulness questionnaire. After completing the questionnaire, participants will be confronted with 7 bowls of granola, each with a different food label. The participant will be asked to choose the most natural granola to eat with the yogurt. After the participant chooses, the participant will then have a selected amount of time to consume the food and then after complete a debrief questionnaire regarding their intake choice. Subjects will be randomized to receive the food items labelled in different orders. The sequences of receiving the food items will be randomly assigned to one of sequences.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65 years' old
* Able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Special dietary patterns that may interfere with study results
* Have allergies/intolerances to foods consumed in the study
* Have uncontrolled high blood pressure at screening visit
* Have uncontrolled elevated fasting blood glucose concentration at screening visit (≥126 mg/dL)
* History of eating disorder
* Planning to become pregnant, pregnant and/or breast-feeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
One choice of 7 Label choices associated with the term 'natural' | 1 hours
  Participant's choice of 7 Label choices associated with the term 'natural'

SECONDARY OUTCOMES:
Amount of Food intake consumption according to label choices | 1 hours
  Amount of Food intake consumption according to label choices

CONTACTS AND LOCATIONS:
Overall Officials: Britt M Burton-Freeman, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No